CLINICAL TRIAL: NCT07251426
Title: Cold atmOspheric plaSMa Therapy Versus standArd Wound Care in Diabetic Foot and Venous Leg ulcerS - a Randomized Controlled Trial
Brief Title: Cold atmOspheric plaSMa Therapy Versus standArd Wound Care in Diabetic Foot and Venous Leg ulcerS
Acronym: COSMAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olaf Bakker (Other)
Responsible Party: Sponsor-Investigator, Olaf Bakker, Principal Investigator, St. Antonius Hospital
Organization: St. Antonius Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL009805; NL009805 (Other: COSMAS)
Record Dates: First submitted 2025-11-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcer; Venous Leg Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold atmospheric Plasma (Experimental): Cold Atmospheric Plasma Treatment 2x per week
  Interventions: Device: COLD ATMOSPHERIC PLASMA
- Standard Wound Care (No Intervention): The use of standardized wound care 2x per week

INTERVENTIONS:
Device: COLD ATMOSPHERIC PLASMA — Cold Atmospheric plasma treatment in addition to standard wound care
  Arms: Cold atmospheric Plasma

SUMMARY:
Chronic wounds such as diabetic foot ulcers (DFUs) and venous leg ulcers (VLUs) pose a major health burden to the patients but also to the healthcare system because of their distorted healing capacity. This is mainly due to a prolonged treatment duration, high recurrence rates and substantial healthcare costs in wound care. Current guidelines exist that outline the standard wound care (SWC) in these patient groups but it often fails to achieve timely healing. Cold atmospheric plasma (CAP) is an emerging technology with promising antimicrobial and wound healing properties. In vitro and in vivo studies have highlighted the ability of CAP to reduce the bacterial biofilm load and stimulate tissue regeneration and microcirculation. This Randomized Controlled Trial (RCT) aims to evaluate the clinical effectiveness and cost-effectiveness of CAP in addition to SWC in patients with a DFU and VLU.

ELIGIBILITY:
Inclusion Criteria:

* 1. is referred to one of the participating hospitals for treatment of a diabetic foot ulcer (DFU) or venous leg ulcer (VLU) with healing stagnation and

  a. For VLU: i. An ulcer on the lower leg resulting from malfunctioning venous valves in the leg veins.

  b. For DFU: i. An ulcer on the foot or lower leg in person with currently or previously diagnosed diabetes mellitus and usually accompanied by neuropathy and/or peripheral artery disease (PAD) in the lower extremity Note: In patients with both diabetes and chronic venous insufficiency, ulcers will be categorized as DFU in case of symptoms of diabetic neuropathy or loss of protective sensation, and otherwise categorized as VLU.

  2. has a wound with a minimum wound surface area of 0.5 cm2 and a maximum diameter of 6 cm (~28 cm2 wound surface area for circular wounds; measured after debridement),

  3. has a minimum age of 18 years old.

Exclusion Criteria:

* 1. the participant has one or more of the following contraindications for PLASOMA:

  1. extreme exudative wounds, i.e. wounds in which moisture is visible within seconds after patting dry;
  2. any implanted active electronic device, such as a pacemaker, is present;
  3. an electronic medical device attached to the body, for example electronic life support equipment, a hearing aid, insulin pump or dialysis machine. If this medical device can be disconnected, PLASOMA treatment may be performed. If the sole purpose of this medical device is monitoring, such as a glucose sensor, PLASOMA treatment is not contra-indicated but note that use of PLASOMA together with such devices has not been tested and may lead to erroneous operation of the attached device during PLASOMA treatment;
  4. metal in the area 10 cm around pad-electrode area, e.g. metal sutures and implants;
  5. connection from outside the body to (near) the heart is present, e.g. a central venous catheter;
  6. the participant has epilepsy;
  7. the participant is pregnant.

     2. the participant has more than one wound that requires professional wound care.

     3. for DFU the WIfI-classification is wound grade 3, defined as an extensive, deep ulcer involving forefoot and/or midfoot; deep, full thickness heel ulcer + calcaneal involvement.

     4. presence of ischemia grade 2 or 3, according to the WIfI classification (= the ankle-brachial pressure index (ABI) is ≤0.59 OR the ankle systolic pressure is ≤69 mmHg OR the toe pressure is ≤39 mmHg; there should be at least one of these three measurements available).

     5. a deep infection defined as an infection of the wound involving structures deeper than skin and subcutaneous tissues (e.g., abscess, osteomyelitis, septic arthritis, fasciitis).

     6. the wound is located on a toe.

     7. the participant receives treatment with immunosuppressive agents or oral corticosteroids; no exclusion if participant has received a stable dose for at least 2 months and the oral corticosteroid dose does not exceed 7.5 mg/day prednisone or equivalent.

     8. the participant is receiving or likely to receive offloading with a total contact cast or advanced wound therapies - such as negative pressure therapy, hyperbaric oxygen therapy, biologicals (e.g. skin substitutes, growth factors), electrophysical therapy - for the to be-treated wound. Advanced wound dressings (including but not limited to hydrocolloid, hydrogel, alginate, collagen and antimicrobial dressings) are not excluded.

     9. presence of a chronic or active skin disorder that may negatively influence wound healing (such as Marfan or Ehlers-Danlos syndrome).

     10. the participant takes part in another study that is likely to compromise the outcome of this study or the feasibility of the participant fulfilling this study.

     11. the participant is lactating.

     12. the participant is unable to provide consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 494 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer-free survival days | 26 weeks
  number of days within the follow-up period (until 26 weeks after the start of the treatment) where the participant is alive and has no ulcer on the same anatomical location of the same foot or limb

SECONDARY OUTCOMES:
Quality of Life (QoL) | baseline, 13 weeks and 26 weeks
  The quality of life will be determined using the questionnaires EQ-5D-5L (generic). EQ-5D-5L descriptive system is divided into five levels of perceived problems: mobility, self-care, usual activities, pain/discomfort, anxiety/depression.
  LEVEL 1: no problem LEVEL 2: slight problems LEVEL 3: moderate problems LEVEL 4: severe problems LEVEL 5: unable to/extreme problems Best outcome is therefore a score of 1 in all categories (total score=5), and worst outcome is a score of 5 in all categories (total score=25).
Wound Quality of Life (Wound-QoL) | baseline, 13 weeks, 26 weeks
  The wound-QoL (wound-specific Quality of Life) will also be measured since complex wounds have a major impact on patients' well-being. The questionnaire is made of three subscales, body, psyche and everyday life. Answers to each item are coded with numbers (0='not at all' to 4='very much'). Minimal score is therefore 0 (no impairement) and maximal 17 (maximum impairement). The higher the outcome the worst the quality of life.
Wound healing rate | 26 weeks
  is defined as the percentage of wounds that are healed
time to wound healing | 26 weeks
  defined as the period measured in days between the start of the treatment period and confirmed wound healing as defined under primary endpoint
Surface area reduction | 26 weeks
  defined as the percentage of wound area reduction, measured using the eKare insight app, which automatically measures the wound metrics. Surface area reduction can show the added value for wounds that are not healed
Recurrences | 26 weeks
  presence of an ulcer at the same anatomical location of the same foot or limb of the initially treated ulcer
Development of new ulcers | 26 weeks
  defined as a new break in the skin not classified as a recurrence, thus not on the same location as the initially treated ulcer
Wound pain | 26 weeks
  Chronic wound pain level is evaluated using question 1 of the Wound-QoL (quality of life) questionnaire to identify any reduction in wound pain. Answers are coded with numbers (0='not at all' to 4='very much'). Minimal score is therefore 0 (no impairement) and maximal 4 (maximum impairement). The higher the outcome the worst the pain level.
Wound infection | 26 weeks
  the percentage wound infections is another measure of treatment efficacy, as CAP is bactericidal, and may indicate potential for reduction in use of antibiotics
Occurence of adverse events | 26 weeks
  will be recorded according to article 80 of the Medical Device Regulation
presence of amputations | 26 weeks
  presence of amputations on the same limb as the treated ulcer, occurring during the treatment or follow-up period (classified as yes/no).
Cost of Care | 26 weeks
  the total healthcare costs related to the treatment of the ulcer during the treatment and follow-up period, including the costs of wound care materials, healthcare professional time, hospital visits, interventions and other medical resource use
Cost Effectiveness | 26 weeks
  the cost per unit of clinical benefit evaluated by comparing the total costs between the intervention and control group in relation to the primary outcome

IPD SHARING:
Plan to Share IPD: Undecided